CLINICAL TRIAL: NCT00219700
Title: Phase II, Randomized, Blinded Study of Ibuprofen-PC and Ibuprofen in Patients With Osteoarthritis to Investigate Efficacy and Gastrointestinal Toxicity
Brief Title: Ibuprofen-PC Compared With Ibuprofen in a GI Safety Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Texas Higher Education Coordinating Board (Other Government)
Responsible Party: Ron Zimmerman/President, PLx Pharma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PL-IB-002
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-11

CONDITIONS: Osteoarthritis
Keywords: NSAID-PC; IBU-PC
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ibuprofen-PC

SUMMARY:
To determine the safety and efficacy of 3 x 800 mg/day IBU-PC assessed by endoscopy and incidence of adverse events

ELIGIBILITY:
Inclusion Criteria:

* moderate osteoarthritis in the hip and/or knee requiring chronic pain medication
* others per protocol

Exclusion Criteria:

* sensitivity to NSAIDs and lecithin
* hypertension
* history of GI and other specific problems
* use of medications and other criteria per the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2005-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Lanza score assessed by endoscopy at baseline and after six weeks of treatment to measure GI safety.

SECONDARY OUTCOMES:
WOMAC and VAS scores every two weeks until end of treatment to measure efficacy.